CLINICAL TRIAL: NCT03540251
Title: Auricular Points Sticking for the Treatment of Hot Flashes in Breast Cancer Patients, a Randomized, Controlled Trial
Brief Title: Clinical Study on Auricular Points Sticking Plus Chinese Medication for Hot Flashes in Breast Cancer Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Longhua Hospital (Other)
Responsible Party: Principal Investigator, Sheng Liu, professor, Longhua Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LonghuaH
Record Dates: First submitted 2018-02-10; First posted 2018-05-30 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer; Hormonal Therapy; Hot Flashes; Acupuncture
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic auricular points treatment (Active Comparator): Therapeutic auricular points treatment including auricular points:CO18、TF2、TF4、AT4、CO15（with complaint of sweating）or CO12(with symptom of heart palpitation)in accordance with the position of auricular points Location map of national standard(GBVT13734-2008) Both groups received a booklet with information about self-care indications, auricular points and its management, and patients can record their hot flash score each day for 12 weeks in the booklets. In addition, both group received 8 treatment sessions of sticking and pressing predefined auricular points.
  Interventions: Other: Auricular Points Sticking
- Placebo auricular points treatment (Sham Comparator): Placebo auricular points treatment including auricular points AH9、AH11、TG3、AT2、LO4 in accordance with the position of auricular points Location map of national standard(GBVT13734-2008) Both groups received a booklet with information about self-care indications, auricular points and its management, and patients can record their hot flash score each day for 12 weeks in the booklets.In addition, both group received 8 treatment sessions of sticking and pressing placebo auricular points treatments.
  Interventions: Other: Auricular Points Sticking

INTERVENTIONS:
Other: Auricular Points Sticking — Auricular Points Sticking is a kind of acupunture based on Meridians Theory of traditional Chinese Medicine.Sticking and pressing predefined therapeutic auricular points can relieve the frequency and severity of hot flashes and other climacteric symptoms.
  Both groups received a booklet with information about self-care indications, auricular points and its management, and patients can record their hot flash score each day for 12 weeks in the booklets.In addition, both group received 8 treatment sessions of sticking and pressing predefined auricular points or placebo auricular points treatments.

SUMMARY:
Object:The aim of this study was to investigate the effectiveness of sticking and massaging auricular points for the management of hot flashes in postoperative breast cancer patients.

DETAILED DESCRIPTION:
Patients and Methods A randomized controlled trial is conducted by comparing effectiveness of sticking and massaging auricular points relieving hot flashes in women with breast cancer versus placebo auricular points. A total of 92 women(still recuiting) with breast cancer, who were under hormonal therapy were randomly assigned and the allocation ratio was 1:1. Both groups received a booklet with information about self-care indications, auricular points and its management, and patients can record their hot flash score each day for 12 weeks in the booklets.In addition, both group received 8 treatment sessions of sticking and pressing predefined auricular points or placebo auricular points treatments.

The primary outcome was hot flash score(HFS)at the end of treatment (week 12), calculated as the frequency multiplied by the average severity of hot flashes.The secondary outcomes were climacteric symptoms and quality of life, measured by the Greene Climacteric Scale(GCS)and Menopause Quality of Life scales(MenQoL)as well as serum estradiol(E2), follicle-stimulating hormone(FSH) and beta-endorphin(β-EP).Expectation and satisfaction of treatment effect and safety were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer after surgical treatment, pathologically diagnosed malignant breast epithelial tumors (breast cancer), immunohistochemistry showed pathological type of estrogen receptor (ER) and / or progesterone receptor (PR) positive.
* Participants should be currently receiving endocrine therapy with oral administration of SERMS(selective estrogen receptor modulators) only.
* Participants should be suffered from perimenopausal symptoms,which is the sudden onset of facial skin flushing, sweating, began from chest and neck,often lasts a few seconds to several minutes and then subsided after center body temperature drops, the associated symptoms of heart palpitations, anxiety, impatience and even a sense of panic, and even wake up at night. The interval between the two attacks is more than 10 minutes.
* Hot flashes occurs during endocrine therapy of breast cancer
* KPS score >60 score >2 and ECOG
* Hot flashes (greater than or equal to 3 times the number of hot flashes per day)
* Symptoms persist for more than 2 weeks

Exclusion Criteria:

* Participants who have uncontrolled diabetes, hyperthyroidism and hypertension and in patients with pheochromocytoma
* Abnormal blood routine, liver and kidney damage (the index is greater than 1.2 times the upper limit of normal value)
* Pregnant or lactating women, persons with mental disorders
* Participants with other cancers
* Participants are participating in other clinical trials
* Current chemotherapy treatment period has not yet completed
* Taking corticosteroids or sex hormone treatment.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — postoperative breast cancer patients who are receiving who hormonal therapy
Enrollment: 92 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Hot Flash Score at 12 weeks | "an average of 1 year" Collect all cases and fill in CRFs;"up to 24 weeks"log in data and complete statistics;"up to 24 weeks"refine the paper and publish articles
  Each week's average HFS of both treatment and placebo group was recorded and all the findings were statistically treated by General Estimation Equation(GEE) .

SECONDARY OUTCOMES:
Change from Baseline GCS and MenQoL at 12 weeks | "an average of 1 year" Collect all cases and fill in CRFs;"up to 24 weeks"log in data and complete statistics;"up to 24 weeks"refine the paper and publish articles
  The GCS, also known as Greene Climacteric Scale and MenQoL Score(Menopause-specific Quality of Life Scale) before and after therapy were the secondary outcome measures, the data were statistically analyzed with ne sample t test if conforming to normal distribution, or otherwise, rank tests and Chi-square test should be utilized to analysis the data.
Change from Baseline beta-EP at 12 weeks | "an average of 1 year" Collect all cases and fill in CRFs;"up to 24 weeks"log in data and complete statistics;"up to 24 weeks"refine the paper and publish articles
  The serum beta-EP before and after therapy was another secondary outcome measure, the laboatatory outcomes were also statistically analyzed with one sample t test.

OTHER OUTCOMES:
Safety and Tolerability-treatment-related adverse events | "an average of 1 year" Collect all cases and fill in CRFs;"up to 24 weeks"log in data and complete statistics;"up to 24 weeks"refine the paper and publish articles
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Liu, Doctor, Study Director — Shanghai University of Traditional Chinese Medincine Afflicated Longhua Hospital
Locations (1):
- Longhua Hosptial, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided